CLINICAL TRIAL: NCT03484286
Title: Selfcare Management Intervention in Heart Failure
Acronym: SMART-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Sofia Gerward, Principal Investigator, MD, PhD, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMART-HF
Record Dates: First submitted 2018-03-22; First posted 2018-03-30 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallell randomized clinical trial with continuous sampling and a 1:1 randomization.
Who Masked: Outcomes Assessor
Masking Description: Cardiovascular events will be adjudicated as heart failure related or not.
  Data analysis will be performed by staff blinded to the patients IDs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Subject to standard care. No interventions above and beyond what is deemed standard care for heart failure patients in the region where the study takes place.
  Interventions: Other: Standard care
- Intervention group (Experimental): Device: OPTILOGG
  Interventions: Device: OPTILOGG

INTERVENTIONS:
Device: OPTILOGG — OPTILOGG is a CE marked class 1m medical device. It consists of a tablet computer and a wirelessly connected weight scale. The system will have some patient specific information regarding the flexible (loop-) diuretics scheme.
  The patient will be asked to step on the weight scale daily, and will be shown to some brief information on how to live better with HF, as well as the recommended dose of diuretics that specific day. Every five days the patient will answer three questions about his/her symptoms, namely shortness of breath, fatigue and peripheral edema. The system also contains information that the patient can study at his/her leisure. If the system detects a deterioration in HF status, the patient is encouraged to contact his/her health care provider via telephone.
  Arms: Intervention group
Other: Standard care — Patients in the control group will be subject to standard heart failure care.
  Arms: Control group

SUMMARY:
A novel tool for self-care enhancement for heart failure (HF) patients has been developed. In this randomized controlled trial, patients will be randomized 1:1 to either receive the home-based tool (OPTILOGG) or standard care. The intervention will go on for 8 months, and outcomes are self-care, cardiovascular events (including emergency visits, admissions, number of in-hospital days).

DETAILED DESCRIPTION:
Patients will be recruited using continuous sampling, and will be approached either in connection with being discharged after a heart failure (HF) related event or upon visiting an out-patient HF clinic if the patient has been admitted for HF at least once the last year.

After written consent has been given, demographical data will be noted, and the patient will complete forms: the European Heart Failure Self-care Behaviour scale 9-item questionnaire (EHFScB-9) and self-assessment of symtoms (NYHAclass). Expected time for this is 20 minutes. The baseline demographical data will include age, gender, ejection-fraction, New York Heart Association (NYHA)-class, blood pressure, heart rate, HF aetiology, and other routine tests for HF visits as outlined in the European guidelines for HF treatment.

After the patient has filled out the forms, the patient will be randomized to the control group (CG) meaning standard care, or the intervention group (IG). Patients allocated to the IG will be equipped with the home based self-care enhancement tool OPTILOGG. OPTILOGG assists the patient with symptom monitoring and flexible diuretics regimen, as well as education about living with HF. It consists of a specialized tablet computer wirelessly connected to a weight scale. OPTILOGG is CE-marked. The intervention will be deployed for eight months. After the eight months, the patients will be called to a follow-up visit. During the visit all data that was collected at baseline/recruitment will be collected again. All cardiovascular events for each patient will be retrieved, for the eight months during which the intervention was deployed, but also for the following 12 months. These events include hospital admissions, ER-visits and number of in-hospital days.

Based off of previous findings in the literature, target for enrollment was set at 70 + 70 patients, to achieve statistical significance with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed heart failure, International classification of diseases (ICD): I50, existing or de-novo, in NYHA-class II-IV
* Admission for HF within the last 12 months
* Filled out consent form
* Expected to be able to use the tool, if allocated to the intervention group

Exclusion Criteria:

* Decline to participate
* More than mild cognitive impairment
* Expectancy of life < 8 months
* For other reasons deemed inappropriate to be enrolled, e.g. participating in another study affecting standard care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Self-care behaviour | Eight months
  Registered using the European Heart Failure Self-care Behaviour Scale (EHFScB), a validated instrument for measuring heart failure (HF) self-care behaviour. The questionnaire is made up of 9 items, where the respondent can choose between 5 different answers to each of the 9 statements. Each item thus generates a score between 1 and 5. The total score for the instrument is between 9 and 45, with 9 constituting the best, or most desireable self-care behaviour and 45 the worst.
  Data will be analyzed on a group level using Mann-Whitney-U test for independent samples.

SECONDARY OUTCOMES:
Number of HF related days in the hospital | Eight months
  All in-hospital days will be adjudicated as HF-related, or non-HF related. The HF-related in-hospital days will then be analyzed on the group level.
Event-free survival | Eight months
  Composite endpoint of HF-admissions, HF related ER visits, all-cause mortality

OTHER OUTCOMES:
Number of HF admissions | Eight months
  All admissions will be adjudicated as HF-related or non-HF related, and the frequency of hospital admissions for HF will be analyzed on the group level.
Number of ER-visits | Eight months
  It is possible that patients get admitted through other pathways than through the ER. To analyze this we will analyze HF-related ER-visits and contrast with HF-admissions to explore potential differences in care pathways between the two groups.
Adherence to the intervention | Eight months.
  Each system will register all patient interactions. The adherence for each patient expressed as a frequency will be analyzed. This only pertains to the IG.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Gerward, PhD, Principal Investigator — Lund University
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No